CLINICAL TRIAL: NCT04966078
Title: Comparison Between Liposuction and Peri-areolar Surgical Excision in Mild and Moderate Cases of Gynaecomastia
Brief Title: Treatment of Mild and Moderate Cases of Gynaecomastia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Diaa eldeen abd elraheem mohamed, principal investigator, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-21-07-10
Record Dates: First submitted 2021-07-13; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Gynecomastia
MeSH Terms: conditions — Gynecomastia | interventions — Lipectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- liposuction (Active Comparator): group A will be treated with liposuction
  Interventions: Procedure: liposuction
- periareolar surgical excision (Active Comparator): Group B will be treated with periareolar surgical excision
  Interventions: Procedure: surgical excision

INTERVENTIONS:
Procedure: liposuction — suction-assisted liposuction
  Arms: liposuction
Procedure: surgical excision — periareolar surgical excision
  Arms: periareolar surgical excision

SUMMARY:
This study aims to compare liposuction and periareolar surgical excision in mild and moderate cases of gynecomastia as regard cosmosis, complications, patient satisfaction, operation time, and hospital stay.

This study will be carried out on patients with gynecomastia presented to the Plastic Surgery Department, Sohag University, in the period between January 2021 to January 2022 as a retrospective and prospective study.

Patients will be divided into 2 groups:

group A treated with suction-assisted liposuction. group B treated with peri-areolar surgical excision. Each group contains 20 patients.

ELIGIBILITY:
Inclusion Criteria:

- The age of patients ranges from 18-60yrs. Mild and moderate cases of gynecomastia.

Exclusion Criteria:

* Patients with endocrine causes. Patients with genetic causes. Severe cases of gynecomastia. Patients who refused surgical intervention. Patients who are not fit for surgery. Patients with chronic illness.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Difference between group A and B in aesthetic satisfaction | difference between group A and B in aesthetic results according to visual analogue scale at 3 month post-operative
  A 100 -point visual analogue scale (VAS) for the assessment of aesthetic satisfaction with 0 as the worst cosmosis and 100 as the best aesthetic result With filled standardized charts.

CONTACTS AND LOCATIONS:
Overall Officials: Gamal Y Elsaied, MD, Study Chair — sohag univeristy hospital
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No